CLINICAL TRIAL: NCT04599582
Title: Prospective Randomised Study of a New Anteverted Uncemented Stem. Randomised Study Between the SP-CL and the Corail Stem With the Use of a Delta Cup.
Brief Title: Prospective Randomised Study of a New an Uncemented Stem.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Link America, Inc. (Industry)
Responsible Party: Principal Investigator, Johan Karrholm, Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kärrholm: SPCL study
Record Dates: First submitted 2020-10-13; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Hip Osteoarthritis
Keywords: hip arthroplasty; Joint replacement; Uncemented stem; Anatomical stem
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SP-CL (Active Comparator)
  Interventions: Device: Hip Arthroplasty
- Corail (Active Comparator)
  Interventions: Device: Hip Arthroplasty

INTERVENTIONS:
Device: Hip Arthroplasty — Patients are operated with hip replacement.

SUMMARY:
Patients will be randomised to either operation with a Corail stem or a SP-CL stem. The groups are examined with RSA, conventional x-rays, PROM-data and DXA. First evaluation will be done at two years.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoartritis Secondary osteoartritis

Exclusion Criteria:

* Ongoing treatment with corticoid steroids, Active cancer disease, previously known osteoporosis or osteomalacia, inflammatory arthritis, unsuitable anatomy, difficulties to speak or understand the Swedish language.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Oxford hip score | two years
  Patient reported outcome measure

SECONDARY OUTCOMES:
RSA-examination | two years
  Migration of stem
Conventional X-rays | two years
  Detection of radiolucent lines
Harris hip score | two years
  Patient reported outcome
DXA | Two years
  Change of bone mineral density

IPD SHARING:
Plan to Share IPD: No